CLINICAL TRIAL: NCT04282603
Title: Nutritional Strategies for Metabolic Health in Aging
Acronym: NSMH
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Grant Transfer Not Approved
Sponsor: University of Alaska Fairbanks (Other)
Responsible Party: Principal Investigator, Robert "Trey" H. Coker, Professor of Biology, University of Alaska Fairbanks
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1427567-2
Record Dates: First submitted 2020-02-05; First posted 2020-02-25 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Sarcopenic Obesity
Keywords: Adipose tissue; Skeletal Muscle; Physical Function

STUDY DESIGN:
Intervention Model Description: The study design is a randomized, double blind, two arm study, where one arm receives a standard meal replacement (Bariatrics Advantage), and the other an enhanced one (ie., EMR) for 24 weeks, including a caloric restriction period of 12 weeks, and a maintenance period of 12 weeks.
Who Masked: Participant, Investigator
Masking Description: Eligible volunteers will be randomly assigned to one of two groups: Experimental Meal Replacement or Bariatrics Advantage Meal Replacement. Only the statistician will know to which group a subject is assigned. Identifying information with regard to randomization of participants to their assigned group will be stored in a binder with Case Report Forms. A master list linking participants to a number and their assigned group will be kept in a password protected file in the database by the study statistician. This process will ensure a high degree of scientific rigor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Meal Replacement (Experimental): Participants randomized to this arm will consume 5 servings/day of experimental meal replacement in conjunction of 400 kcal of solid food for 12 weeks during the weight loss portion of the trial. This will be followed by the consumption of 1 serving/day of experimental meal replacement for 12 weeks during the weight maintenance portion of the trial.
  Interventions: Combination Product: Weight Loss and Weight Maintenance
- Bariatrics Advantage Meal Replacement (Active Comparator): Participants randomized to this arm will consume 5 servings/day of Bariatrics Advantage meal replacement in conjunction of 400 kcal of solid food for 12 weeks during the weight loss portion of the trial. This will be followed by the consumption of 1 serving/day of Bariatrics Advantage meal replacement for 12 weeks during the weight maintenance portion of the trial.
  Interventions: Combination Product: Weight Loss and Weight Maintenance

INTERVENTIONS:
Combination Product: Weight Loss and Weight Maintenance — Participants will consume a 1,200 kcal/day diet for twelve weeks. This is the amount of calories most commonly provided in medical weight loss programs, and considered the maximum allowable caloric intake to induce a physiologically significant weight loss. Following the weight loss portion of the trial, participants will enter the twelve week maintenance period, during which time they will consume one serving per day in place of lunch of the same meal replacement beverage used during medical weight loss.

SUMMARY:
Sarcopenic obesity in older individuals presents a clinical conundrum without an effective therapeutic strategy. This study will determine the impact of precision amino acid delivery as part of a meal replacement (EMR) during weight loss on the preservation of lean tissue and improvements in metabolic health and physical function in older obese adults. Following weight loss, the investigators will examine whether one serving/day of EMR will sustain the above stated benefits.

DETAILED DESCRIPTION:
The health status of the aging population is negatively affected by sarcopenic obesity as described by the progressive loss of lean tissue and an increase in adipose tissue. This condition presents a clinical conundrum as it predisposes older obese individuals to a high risk for disability, morbidity and mortality. Insulin resistance, chronic inflammation, elevations in intrahepatic lipid and detrimental alterations in the gut microbiome are also evident. The application of caloric restriction-induced weight loss (CRWL) used to address these health risks in younger individuals may exacerbate muscle wasting and increase morbidity in older adults. Unfortunately, low fitness levels and poor compliance limit the mitigating influence of weight loss through exercise training on sarcopenic obesity. In order to address anabolic resistance or the decreased ability to maintain protein synthesis that contributes to sarcopenic obesity, the investigators have developed a complete meal replacement that contains a mechanism-targeted profile of essential amino acids (17 grams). This profile is designed to overcome anabolic resistance and maintain net protein balance even in the hypocaloric state. It is our overarching hypothesis that EMR will promote the retention of lean tissue mass, and improve metabolic and functional outcomes following 12 weeks of CRWL, and that those endpoints will be sustained over a 12 week maintenance period with the once per day (q.d.) consumption of EMR. The investigators will randomly assign older obese individuals to either EMR or an isocaloric serving of Bariatrics Advantage (meal replacement that contains 27 grams of intact protein) during these interventions. The investigators will execute these specific aims to test our hypotheses: SA1. Establish the importance of EMR in the preservation of lean tissue mass during CRWL. Lean tissue mass and adipose tissue mass will be determined by dual energy x-ray absorptiometry (DXA) and magnetic resonance imaging/spectroscopy (MRI/MRS) scans. MRI/MRS will be used to measure intrahepatic lipid, and the investigators will evaluate alterations in insulin sensitivity using the HOMA score. The investigators will measure potential changes in gut microbiota in collaboration with Dr. Duddleston at the University of Alaska Anchorage. SA2. Determine the influence of EMR on physical function and increased daily activity during CRWL. Slow walking speed is a strong predictor of morbidity and mortality. The investigators chose the 6-minute walk test to represent the primary endpoint for this aim. The investigators will also determine alterations in gait speed, skeletal muscle power and strength and stair climbing ability, and changes in physical activity using Actigraph GT3X+ devices. SA3. Identify whether EMR q.d. will sustain improvements in body composition, physical function and metabolic parameters over a 12 week, maintenance period following CRWL. Since the preservation of lean tissue mass is directly linked to optimal function and metabolic health, the investigators will measure the influence of EMR q.d. on the indices of metabolic health (ie., intrahepatic lipid, insulin sensitivity) and physical function.

ELIGIBILITY:
Inclusion Criteria:

* 60-80 years of age
* Body mass index of 30-40 kg/m2
* Participants must be capable of understanding the consent process
* Participants must be capable of signing the consent form
* Participants must have access to transportation to the clinic site

Exclusion Criteria:

* Creatinine >1.6
* Serum glutamate pyruvate transaminase >2 times normal
* Resting blood pressure above 160/90 mmHg
* Use of Gemfibrozil
* Use of corticosteroids
* Previously diagnosed diabetes (fasting blood glucose ≥ 126 mg/dl)
* History of kidney or liver disease
* Heart disease as indicated by interventional procedures
* Recent history of alcoholism
* Physical or neurological disorder that would prevent them from completing the functional tests
* Lactose intolerance
* Active cancer within the last two years
* Chronic inflammatory conditions that preclude completion of functional tests

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Lean tissue mass and adipose tissue mass | 24 weeks for each participant
  Lean tissue mass and adipose tissue mass will be determined by dual energy x-ray absorptiometry.
Skeletal muscle | 24 weeks for each participant
  Magnetic resonance imaging scans will be used to measure the cross sectional area of skeletal muscle
Metabolic health | 24 weeks for each participant
  The investigators will evaluate alterations in insulin sensitivity using the HOMA score.
Intrahepatic lipid | 24 weeks for each participant
  Magnetic resonance imaging and spectroscopy scans will be used to measure intrahepatic lipid
Physical function | 24 weeks for each participant
  A 6-minute walk test will be used to assess changes in physical function.
Gut microbiome | 24 weeks for each participant
  Stool kits will be provided with standardized instructions to participants for collection and transportation of stool samples. DNA will be extracted to evaluate alterations in gut microbiota.

SECONDARY OUTCOMES:
Timed step test | 24 weeks for each participant
  This test will be used to evaluate dynamic balance ability. The participant will step and down from a 4 inch bench as quickly as possible 5 times.
Timed floor transfer test | 24 weeks for each participant
  This test will be used to evaluate mobility. While being timed, the participant will start in the standing position, go to the supine position and return to the standing position.
Hand grip test | 24 weeks for each participant
  This test will determine muscle strength. The participant will grip the hand dynamometer and perform three tests, alternating with a brief rest period of 20 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Coker, PhD, Principal Investigator — University of Alaska Fairbanks
Locations (1):
- University of Alaska Fairbanks, Fairbanks, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
Structured de-identified clinical data. Restrictive protocols will be in place for human data and for data, if any, owned by Alaska Native tribes. The PI, Data Manager and Project leader will review data requests using criteria including scientific value, appropriate research plan, protection of participant and community confidentiality, and dissemination plan. All persons working with COBRE human data will have to sign a Confidentiality Agreement, Publication Agreement, and submit proof of current Collaborative IRB Training Initiative (CITI) certification or an equivalent approved by the UAF IRB when appropriate. Data access is generally approved for three years, at which time data sets must be destroyed or the data access approval extended.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code